CLINICAL TRIAL: NCT05995379
Title: Donor Derived Cell-free DNA and Rejection of Kidney Allografts
Status: Completed | Type: Observational
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: ddcfDNA_study001
Record Dates: First submitted 2023-07-28; First posted 2023-08-16 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Kidney Rejection Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation cohort
  Interventions: Diagnostic Test: Donor-derived cell-free DNA
- Validation cohort
  Interventions: Diagnostic Test: Donor-derived cell-free DNA

INTERVENTIONS:
Diagnostic Test: Donor-derived cell-free DNA — Cell-free DNA (cfDNA) is fragmented extracellular DNA released in the bloodstream from cells undergoing apoptosis or necrosis. In transplantation, donor-derived cfDNA (dd-cfDNA) is detected in the blood of kidney recipients and has been proposed as a noninvasive biomarker to detect rejection.
  One additional blood sample will be collected and dd-cfDNA levels will be centrally analyzed.

SUMMARY:
To assess the association of dd-cfDNA with the presence, activity and severity of allograft rejection, and determine whether dd-cfDNA adds value to standard of care monitoring parameters in detecting kidney allograft rejection.

ELIGIBILITY:
Inclusion Criteria:

* Recipients transplanted from a deceased or living donor, who undergone a kidney allograft biopsy with clinical, biological, histological and immunological data.
* Written informed consent at the time of transplantation for the center database

Exclusion Criteria:

* Combined organ transplantation
* Pregnant women
* Bone marrow transplant

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Kidney transplant recipients recruited in 14 French centers
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2011-09-21 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
The occurrence of biopsy-proven allograft rejection at the time of dd-cfDNA measurement | The allograft biopsies will be performed at 3 months and 1 year after transplant and/or in for cause biopsies performed at any time post transplantation in unstable patients.
  Biopsy-proven rejection refers to the confirmation of rejection through the examination of kidney allograft tissue obtained from a biopsy procedure. This includes different types of rejection, which are antibody-mediated rejection, T-cell-mediated rejection, and mixed rejection. All the allograft biopsies will be classified according to the most recognized classification (Banff 2019 classification), which provides standardized criteria for the diagnosis and the characterization of the different types of rejection.
  To evaluate the association between dd-cfDNA and the occurrence of rejection, measurement of dd-cfDNA will be done at the time of each biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, Principal Investigator — Paris Institute for Transplantation and Organ Regeneration

REFERENCES:
- [Derived] Aubert O, Ursule-Dufait C, Brousse R, Gueguen J, Racape M, Raynaud M, Van Loon E, Pagliazzi A, Huang E, Jordan SC, Chavin KD, Gupta G, Kumar D, Alhamad T, Anand S, Sanchez-Garcia J, Abdalla BA, Hogan J, Garro R, Dadhania DM, Jain P, Mandelbrot DA, Naesens M, Dandamudi R, Dharnidharka VR, Anglicheau D, Lefaucheur C, Loupy A. Cell-free DNA for the detection of kidney allograft rejection. Nat Med. 2024 Aug;30(8):2320-2327. doi: 10.1038/s41591-024-03087-3. Epub 2024 Jun 2. PMID 38824959

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT05995379/Prot_SAP_000.pdf